CLINICAL TRIAL: NCT03813758
Title: Inter-observer and Intra-observer Variability of the Wrinkle Test and the Optimum Time Need for the Test. Pilot Study
Brief Title: Inter-observer and Intra-observer Variability of the Wrinkle Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, guy rubin, MD, HaEmek Medical Center, Israel
Other Study IDs: 134-18-EMC
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Wrinkle Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- finger after digital nerve cut
  Interventions: Diagnostic Test: wrinkle test
- healthy finger
  Interventions: Diagnostic Test: wrinkle test

INTERVENTIONS:
Diagnostic Test: wrinkle test — soaking in 40 deg water for 40 min. every 10 min the hand will be photo

SUMMARY:
Skin wrinkling of the fingers following immersion in warm water depends on intact sympathetic innervation. It is abolished by lesions affecting both central and peripheral sympathetic pathways. It affords a simple and reliable clinical test of sympathetic function.

DETAILED DESCRIPTION:
Fingertip skin wrinkling after prolonged immersion in water is a well-recognized phenomenon, whereas a denervated digit does not exhibit normal skin wrinkling while a finger with a regenerated or repaired nerve shows at least partial reappearance of wrinkling. This is the basis for the bedside immersion-wrinkling test of autonomic digital nerve function. The exact mechanism of fingertip skin wrinkling is still subject to controversy. the purpose of this study is to examine the Inter-observer and Intra-observer Variability of the Wrinkle Test.

ELIGIBILITY:
Inclusion Criteria:

* patients after suture of full cut of digital nerve

Exclusion Criteria:

* other nerve injury

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients after suture of full cut of digital nerve
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
wrinkle test | 40 min
  wrinkle of the skin in the finger compaared to the finger witout digital nerve injury

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No